CLINICAL TRIAL: NCT00264303
Title: A Comparative Study on Clinical Efficacy and Safety of Levocetirizine 5 mg Oral Capsules Once Daily in the Morning vs. Desloratadine 5 mg Oral Capsules Once Daily in the Morning in Patients Suffering From Chronic Idiopathic Urticaria (CIU)
Brief Title: CUTE (Chronic Urticaria Treatment Evaluation)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00394; EudraCT 2005-000358-65; CUTE
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Idiopathic Urticaria
Keywords: Chronic Idiopathic Urticaria; CUTE Levocetirizine Xyzal®
MeSH Terms: conditions — Chronic Urticaria | interventions — levocetirizine; desloratadine

ARMS (2):
- Levocetirizine (Experimental): Levocetirizine, once daily, 4 week duration
  Interventions: Drug: Levocetirizine
- Desloratadine (Active Comparator): Desloratadine, once daily, 4 week duration
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Levocetirizine — 5mg oral capsules, once daily, 4 week duration
  Arms: Levocetirizine
Drug: Desloratadine — 5mg oral capsules, once daily, 4 week duration
  Arms: Desloratadine

SUMMARY:
A study to compare the clinical efficacy and safety of Levocetirizine vs. Desloratadine in patients suffering from Chronic Idiopathic Urticaria (CIU) measured by the mean pruritus severity score over the first week of treatment

ELIGIBILITY:
Inclusion Criteria:

- At visit 1: Clinical history of Chronic Idiopathic Urticaria for a period of at least 6 weeks during the last 3 months without an identifiable cause

- At visit 2 (after a baseline period of at least 3 days): patient with adequate signs of CIU, both in terms of symptoms and severity.

Exclusion Criteria:

- Any condition that would interfere with the evaluation of the therapeutic response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 886 (Actual)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (80):
- Belgium (6):
  - Bruges
  - Brussels
  - Liège
  - Merksem
  - Sint-Niklaas
  - Woluwe-St-Lamb
- France (17):
  - Bernay
  - Besançon
  - Hyères
  - Les Milles
  - Marseille
  - Montpellier
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Poitiers
  - Quimper
  - Saint-Mandé
  - Troyes
  - Valence
  - Villejuif
- Germany (14):
  - Augsburg
  - Berlin
  - Cologne
  - Dresden
  - Düsseldorf
  - Erlangen
  - Göttingen
  - Hamburg
  - Hanover
  - Leipzig
  - Mahlow
  - Mainz
  - München
  - Viersen
- Italy (11):
  - Caserta
  - Catania
  - Cesena
  - Genova
  - Modena
  - Palermo
  - Pavia
  - Roma
  - Siena
  - Udine
  - Verona
- Malaysia (7):
  - Johor Bharu
  - Kelantan
  - Kuala Lumpur
  - Negeri Sembilan
  - Perak
  - Pulau Pinang
  - Sarawak
- Romania (4):
  - Brasov
  - Bucharest
  - Dolj
  - Sibiu
- South Africa (3):
  - Cape Town
  - Durban
  - Lenasia
- Spain (11):
  - A Coruña
  - Albacete
  - Barcelona
  - Granada
  - Madrid
  - Málaga
  - Murcia (El Palmar)
  - Oviedo
  - Santiago de Compostela
  - Seville
  - Valencia
- United Kingdom (7):
  - Amersham
  - Cardiff
  - Irvine
  - Leicester
  - London
  - Nuneaton
  - Salford

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 976 patients have been screened for this study. Ninety patients were ineligible for randomization, 886 have been randomized and treated. Participants flow and Baseline Characteristics refer to all patients randomized and treated.
Groups:
- Levocetirizine 5 mg: Levocetirizine 5 mg once daily for four weeks
- Desloratadine 5 mg: Desloratadine 5 mg once daily for four weeks
Period: Overall Study
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Started | 438 | 448
Completed | 413 | 419
Not Completed | 25 | 29
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 10 | 13
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Various reasons listed in study report | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg | Total
Number analyzed (Participants) | 438 | 448 | 886
Age Continuous [Mean (Standard Deviation); unit: years] | 43.4 (15.3) | 42.9 (14.9) | 43.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 306 | 590
  Male | 154 | 142 | 296
Region of Enrollment [Number; unit: participants]
  France | 79 | 82 | 161
  Malaysia | 45 | 44 | 89
  Spain | 38 | 37 | 75
  Belgium | 14 | 10 | 24
  Romania | 57 | 56 | 113
  South Africa | 30 | 30 | 60
  Germany | 109 | 115 | 224
  Italy | 62 | 65 | 127
  United Kingdom | 4 | 9 | 13

OUTCOME MEASURES:

1. Secondary Outcome: Mean Chronic Idiopathic Urticaria (CIU) Composite Score Over the First Week of Treatment
Description: CIU composite score is defined as the sum of 2 scores defined on an ordinal 4-point scale (pruritus severity score: 0=none, 1=mild, 2=moderate, 3=severe/intense; score for the number of wheals/24 h: 0=none, 1=mild or <=20 wheals, 2=moderate or 21-50 wheals/24 h, 3=severe/intense or >50 wheals/24 h). Mean is averaged over the 1st week of treatment.
Time Frame: over the first week of treatment
Population: Intent to treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 443
Units on a scale | 1.98 (0.08) | 2.23 (0.08)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; Test type: Superiority or Other; p = 0.005, ANCOVA; ANCOVA with treatment and pooled center as factors and baseline CIU composite score as covariate; Mean Difference (Net) = 0.25, 95% CI [0.08 to 0.43]

2. Secondary Outcome: Mean Chronic Idiopathic Urticaria (CIU) Composite Score Over the Four Weeks of Treatment
Description: CIU composite score is defined as the sum of two scores defined on an ordinal 4-point scale (pruritus severity score: 0=none, 1=mild, 2=moderate, 3=severe/intense; score for the number of wheals/24 h: 0=none, 1=mild or <=20 wheals, 2=moderate or 21-50 wheals/24 h, 3=severe/intense or >50 wheals/24 h). Mean is averaged over the 4 weeks of treatment.
Time Frame: over the four weeks of treatment
Population: Intent to treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 443
Units on a scale | 1.71 (0.07) | 1.88 (0.07)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; Test type: Superiority or Other; p = 0.041, ANCOVA; ANCOVA with treatment and pooled center as factors and baseline CIU composite score as covariate; Mean Difference (Net) = 0.17, 95% CI [0.01 to 0.34]

3. Secondary Outcome: Mean Pruritus Severity Score Over the Four Weeks of Treatment
Description: Pruritus severity is evaluated on an ordinal 4-point scale from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe/intense). Mean pruritus severity score is averaged over the four weeks of treatment.
Time Frame: over the four weeks of treatment
Population: Intent to treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 443
Units on a scale | 0.86 (0.04) | 0.99 (0.04)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; Test type: Superiority or Other; p = 0.004, ANCOVA; ANCOVA with treatment and pooled center as factors and baseline pruritus severity score as covariate; Mean Difference (Net) = 0.13, 95% CI [0.04 to 0.22]

4. Secondary Outcome: Mean Score for Pruritus Duration Over the First Week of Treatment
Description: The pruritus duration score is evaluated on an ordinal 4-point scale (0=no pruritus, 1=less than 1 hour, 2=1 to 6 hours, 3=more than 6 hours). Mean score for pruritus duration is averaged over the first week of treatment.
Time Frame: over the first week of treatment
Population: Intent to treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 443
Units on a scale | 1.08 (0.04) | 1.24 (0.04)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA with treatment and pooled center as factors and baseline pruritus duration as covariate; Mean Difference (Net) = 0.16, 95% CI [0.06 to 0.26]

5. Secondary Outcome: Mean Score for Pruritus Duration Over the Four Weeks of Treatment
Description: The pruritus duration score is evaluated on an ordinal 4-point scale (0=no pruritus, 1=less than 1 hour, 2=1 to 6 hours, 3=more than 6 hours). Mean score for pruritus duration is averaged over the four weeks of treatment.
Time Frame: over the four weeks of treatment
Population: Intent to treat (ITT) Population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 444
Units on a scale | 0.93 (0.04) | 1.05 (0.04)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; Test type: Superiority or Other; p = 0.009, ANCOVA; ANCOVA with treatment and pooled centers as factors and baseline pruritus duration score as covariate; Mean Difference (Net) = 0.12, 95% CI [0.03 to 0.22]

6. Primary Outcome: Mean Pruritus Severity Score Over the First Week of Treatment
Description: Pruritus severity is evaluated on an ordinal 4-point scale from 0 to 3 (0=none, 1=mild, 2=moderate). Mean pruritus severity score is averaged over the first week of treatment.
Time Frame: over the first week of treatment
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Number analyzed (Participants) | 434 | 443
Units on a scale | 1.02 (0.04) | 1.18 (0.04)
Statistical Analysis 1: Comparison: Levocetirizine 5 mg vs Desloratadine 5 mg; The primary hypothesis to be tested in this study was that the clinical efficacy of Levocetirizine 5 mg is superior to that of Desloratidine 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment and pooled center as factors and baseline severity as covariate; Mean Difference (Net) = 0.16, 95% CI [0.07 to 0.26]

ADVERSE EVENTS:
Arm/Group | Levocetirizine 5 mg | Desloratadine 5 mg
Serious Adverse Events (participants affected / at risk) | 0/438 | 2/448
Other Adverse Events (participants affected / at risk) | 80/438 | 77/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levocetirizine 5 mg (N=438) | Desloratadine 5 mg (N=448)
Diabetes Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levocetirizine 5 mg (N=438) | Desloratadine 5 mg (N=448)
Abdominal pain upper (Gastrointestinal disorders) | 10 | 11
Fatigue (General disorders) | 19 | 14
Headache (Nervous system disorders) | 35 | 48
Nausea (Gastrointestinal disorders) | 5 | 10
Somnolence (Nervous system disorders) | 31 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.